CLINICAL TRIAL: NCT00055224
Title: Predictability and Aversive Expectancies in Anxiety and Depressive Disorders
Brief Title: Expectation of Unpleasant Events in Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 030093; 03-M-0093
Record Dates: First submitted 2003-02-21; First posted 2003-02-21 (Estimated); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2022-08

CONDITIONS: Anxiety Disorders
Keywords: Anxiety Disorder; Psychophysiology; Shock Threat; Context Conditioning; Agoraphobia; Panic Disorder; Generalized Anxiety Disorder; GAD; Healthy Volunteer; HV
MeSH Terms: conditions — Anxiety Disorders; Agoraphobia; Panic Disorder; Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Healthy Participants (Experimental): Substudy 1/ Neutral, Predictable, and Unpredictable Responses (NPU): physiological responses to different threat of shock conditions - no shock, unpredictable shock, and predictable-cued shock. Substudy 2/ Working Memory Task: Subjects performed a working memory task under threat of shock and in safety. Substudy 5 /Face Stroop Task: Stimuli were pictures of faces exhibiting anger, disgust, fear, happiness, sadness, and surprise intermixed with pleasant, unpleasant, and neutral pictures. Substudy 7/ Active Avoidance Signal Task (AAST) and Sustained Attention Response Task (SART): In AAST, participants performed paradigms which tested whether threats impact the initiation and the inhibition of behavioral responses. In SART, participants were presented with stimuli and either initiated a go or nogo response. Pilot Tasks: Participants completed one/more tasks: nerve stimulation, short speech, air burst, saliva samples, squeezer task, virtual reality task, or computer-based task.
  Interventions: Device: Threat of shock
- Anxiety subjects (Experimental): Substudy 1/ Neutral, Predictable, and Unpredictable Responses (NPU): physiological responses to different threat of shock conditions - no shock, unpredictable shock, and predictable-cued shock. Substudy 2/ Working Memory Task: Subjects performed a working memory task under threat of shock and in safety. Substudy 5 /Face Stroop Task: Stimuli were pictures of faces exhibiting anger, disgust, fear, happiness, sadness, and surprise intermixed with pleasant, unpleasant, and neutral pictures. Substudy 7/ Active Avoidance Signal Task (AAST) and Sustained Attention Response Task (SART): In AAST, participants performed paradigms which tested whether threats impact the initiation and the inhibition of behavioral responses. In SART, participants were presented with stimuli and either initiated a go or nogo response. Pilot Tasks: Participants completed one/more tasks: nerve stimulation, short speech, air burst, saliva samples, squeezer task, virtual reality task, or computer-based task.
  Interventions: Device: Threat of shock

INTERVENTIONS:
Device: Threat of shock — During threat, a participant could receive a shock. During safe, a participant could not receive as shock. Participants selected their highest tolerable level of shock.

SUMMARY:
Fear and anxiety are normal responses to a threat. However, anxiety is considered abnormal when the response to the threat is excessive or inappropriate. This study will examine changes in the body and brain that occur during unpleasant learning experiences in healthy volunteers with high, moderate, and low levels of anxiety.

A high degree of generalized anxiety is a component of many anxiety disorders and is regarded as a marker of vulnerability for these disorders. People with anxiety disorders and individuals with high degrees of anxiety have inappropriate expectations of unpleasant events. This study will investigate the development of expecting unpleasant events in healthy volunteers with varying degrees of anxiety using aversive conditioning models. A later phase of the study will enroll participants with anxiety disorders and compare their responses to those of healthy volunteers.

Patients who meet criteria for an anxiety disorder, and healthy volunteers who have no history of psychiatric or major medical illness will be enrolled in this study. Volunteers will come to the NIH Clinical Center three times for outpatient testing....

DETAILED DESCRIPTION:
High-generalized anxiety is a concomitant of many anxiety disorders and is often regarded as a vulnerability marker for these disorders. One characteristic of patients with anxiety disorders and high trait-anxious individuals is inappropriate expectancies of aversive events. The overall aim of the present protocol is to investigate mechanisms that may promote the development of these aversive expectancies using expectancy-based, associative-learning models.

During aversive conditioning in which a phasic explicit-cue (e.g., a light) is repeatedly associated with an aversive unconditioned-stimulus (e.g., a shock), the organism develops fear to the explicit cue as well as to the environmental context in which the experiment took place. We have obtained preliminary evidence suggesting that contextual fear represents aspects of aversive states that are central to anxiety disorders. In this protocol, we seek further evidence for the relevance of contextual fear to mood anxiety disorders.

One important determinant of contextual fear in both humans and animals is predictability: contextual fear increases when aversive events (e.g., electric shock) are unpredictable, as opposed to when they are predictable. The present protocol will examine the role of predictability of aversive states and of conditioning on threat appraisal in individuals with mood and anxiety disorders.

A second aim is to examine the interaction between experimentally-induced anxiety and cognitive processes, more specifically working memory, in mood and anxiety disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Inclusion criteria for both patients and healthy controls

  * All subjects must be able to give written informed consent prior to participation in this study.
  * PATIENTS ONLY: May have DSM-IV-TR diagnoses of an anxiety disorder (GAD; SAD; Panic disorder; specific phobia) or mood disorder (MDD; BP).
  * PATIENTS ONLY: May be taking the mood stabilizers, Depakote or Lithium Carbonate.
  * Speaks English fluently

EXCLUSION CRITERIA:

* Exclusion criteria for healthy subjects

  * Female subjects who are currently pregnant
  * Subjects who meet DSM-IV criteria for current alcohol or substance abuse
  * Subjects with a history of alcohol or substance dependence within 6 months prior to screening
  * Current Axis I psychiatric disorders as identified with the Structured Clinical Interview for DSM-IV-TR axis disorders, non-patient edition (SCID-np). Past history of any psychotic disorder or bipolar disorder.
  * intelligence quotient (I-Q)<80
  * Medical illnesses (such as diabetes or hypertension) or neurological illnesses (such as carpal tunnel syndrome for shocks to be delivered on affected arm; organic brain impairment; seizure disorder) likely to interfere with the study.
  * Subjects who are on a medication that may interfere with the study.
  * Employee of National Institute of Mental Health (NIMH) or an immediate family member who is a NIMH employee.
* Exclusion criteria for patients

  * Patients who would be unable to comply with study procedures or assessments;
  * Female patients who are currently pregnant;
  * Patients who meet DSM-IV criteria for current alcohol or substance abuse
  * Subjects with a history of alcohol or substance dependence within 6 months prior to screening;
  * Patients who are on a medication (other than mood stabilizers lithium carbonate or Depakote) that may interfere with the study
  * Medical illnesses (such as diabetes or hypertension) or neurological illnesses (such as carpal tunnel syndrome; organic brain impairment; seizure disorder) likely to interfere with the study.
  * Patients will be excluded if they have a current or past history of, delirium, dementia, amnestic disorder, any of the pervasive developmental disorders; or cognitive impairment.
  * Current Axis I psychiatric disorders as identified with the Structured Clinical Interview for DSM-IV-TR axis disorders, non-patient edition (SCID) with the exception of the mood and anxiety disorders. Past history of any psychotic disorder or bipolar disorder..
  * IQ<80
  * Employee of NIMH or an immediate family member who is an NIMH employee.
* Additional exclusion criteria for the active avoidance task

  * Color blindness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 921 (Actual)
Dates: Start 2003-03-24 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monique Ernst, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.We plan to only share de-identified data in a repository. No identified data will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be placed into a repository indefinitely. We plan to start uploading data in the next few months and continue until project completion.
Access Criteria: Questionnaire and biophysiological data will be shared into the DSP and repository.

REFERENCES:
- [Background] Grillon C, Ameli R, Goddard A, Woods SW, Davis M. Baseline and fear-potentiated startle in panic disorder patients. Biol Psychiatry. 1994 Apr 1;35(7):431-9. doi: 10.1016/0006-3223(94)90040-x. PMID 8018793
- [Background] Grillon C, Morgan CA 3rd, Davis M, Southwick SM. Effects of experimental context and explicit threat cues on acoustic startle in Vietnam veterans with posttraumatic stress disorder. Biol Psychiatry. 1998 Nov 15;44(10):1027-36. doi: 10.1016/s0006-3223(98)00034-1. PMID 9821567
- [Background] Grillon C, Morgan CA 3rd. Fear-potentiated startle conditioning to explicit and contextual cues in Gulf War veterans with posttraumatic stress disorder. J Abnorm Psychol. 1999 Feb;108(1):134-42. doi: 10.1037//0021-843x.108.1.134. PMID 10066999
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-M-0093.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 921 participants were consented and performed one or more tasks. 3 participated did not perform any study related tasks.
Pre-assignment Details: All sub-studies were conducted at different time points so subjects had the option to participate in multiple sub-studies.
Groups:
- Healthy Participants; Anxiety Subjects: Substudy 1/ Neutral, Predictable, and Unpredictable Responses: This experiment examined physiological responses including startle reflex to different threat of shock conditions (neutral (N)- no shock, unpredictable - shock at any time, and predictable -cued shock (P)). Each of these conditions were signaled by a written text displayed on a computer monitor (e.g., shock only when blue square present).
  Substudy 2/ Working Memory Task: Subjects performed a working memory task in two conditions, under threat of shock and in safety (no threat of shock).
  Substudy 5 /Face Stroop Task: Stimuli were pictures of faces exhibiting anger, disgust, fear, happiness, sadness and surprise. Intermixed with the faces were pleasant, unpleasant, and neutral pictures. Subjects indicated which emotion the face displayed. Accurate response was used as measure of facial emotion recognition.
  Substudy 7/ Active Avoidance and Sustained Attention Tasks: In the active avoidance signal task (AAST), participants performed paradigms which tested whether threat impacts the initiation and the inhibition of behavioral responses. In the sustained attention response task (SART), participants were presented with stimuli and either initiated a response (i.e. "go") or inhibited their response (i.e. "stop") based on what stimuli were presented.
  Pilot Tasks: Participants completed one/more task: nerve stimulation, short speech, air burst, saliva samples, squeezer task, virtual reality task, or computer-based task.
Period: Overall Study Participants
Arm/Group | Healthy Participants | Anxiety Subjects
Started | 557 | 361
Completed | 557 | 361
Not Completed | 0 | 0
Period: Substudy 1
Arm/Group | Healthy Participants | Anxiety Subjects
Started | 23 | 78
Completed | 23 | 78
Not Completed | 0 | 0
Period: Substudy 2
Arm/Group | Healthy Participants | Anxiety Subjects
Started | 42 | 35
Completed | 42 | 35
Not Completed | 0 | 0
Period: Substudy 5
Arm/Group | Healthy Participants | Anxiety Subjects
Started | 33 (Include subjects who previously participated in sub-study 1 (two participants) and sub-study 2 (one participant)) | 36 (Include subjects who previously participated in sub-study 1 (two participants) and sub-study 2 (two participants))
Completed | 33 | 36
Not Completed | 0 | 0
Period: Substudy 7
Arm/Group | Healthy Participants | Anxiety Subjects
Started | 65 (Include subjects who previously participated in sub-study 1 (seven participants), sub-study 2 (1 participant), and sub-study 5 (one participant)) | 91 (Include subjects who previously participated in sub-study 1 (36 participants), sub-study 2 (seven participants), and sub-study 5 (11 participants))
Completed | 65 | 91
Not Completed | 0 | 0
Period: Pilot Tasks
Arm/Group | Healthy Participants | Anxiety Subjects
Started | 406 | 183
Completed | 406 | 183
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Substudy 1/ Neutral, Predictable, and Unpredictable Responses: This experiment examined physiological responses including startle reflex to different threat of shock conditions (neutral (N)- no shock, unpredictable - shock at any time , and predictable -cued shock (P)) in subjects with anxiety disorders and healthy control. Each of these conditions were signaled by a written text displayed on a computer monitor (e.g., shock only when blue square present).
- Substudy 2/Working Memory Task: Subjects performed a working memory task in two conditions, under threat of shock and in safety (no threat of shock). Subjects included participants with anxiety disorder and healthy volunteer.
- Substudy 5/Face Stroop Task: Stimuli were pictures of faces exhibiting anger, disgust, fear, happiness, sadness and surprise (Ekman, 1993). Intermixed with the faces were pleasant, unpleasant, and neutral pictures. Subjects indicated which emotion the face displayed. Accurate response was used as measure of facial emotion recognition. Subjects included participants with anxiety disorder and healthy volunteer.
- Substudy 7/Active Avoidance and Sustained Attention Tasks: In the active avoidance signal task (AAST), participants performed paradigms which tested whether threat impacts the initiation and the inhibition of behavioral responses. In the sustained attention response task (SART), participants were presented with stimuli and either initiated a response (i.e. "go") or inhibited their response (i.e. "stop") based on what stimuli were presented. Subjects included participants with anxiety disorder and healthy volunteer.
- Pilot Task: Participants completed one or more pilot tasks: nerve stimulation, short speech in front of a small audience or in a virtual environment, burst of air to neck, provide saliva samples for cortisol analysis, squeeze a grip device, virtual reality task, and/or computer based experimental tasks.
- Total: Total of all reporting groups
Arm/Group | Substudy 1/ Neutral, Predictable, and Unpredictable Responses | Substudy 2/Working Memory Task | Substudy 5/Face Stroop Task | Substudy 7/Active Avoidance and Sustained Attention Tasks | Pilot Task | Total
Number analyzed (Participants) | 101 | 76 | 62 | 90 | 589 | 918
Age, Categorical [Count of Participants; unit: Participants] — Population: Study comprised of several sub-studies with the aim of comparing Healthy participants to Anxiety participants
  Participants
    Healthy participants: number analyzed (Participants) | 23 | 42 | 30 | 56 | 406 | 557
    Healthy participants: <=18 years | 0 | 0 | 0 | 0 | 0 | 0
    Healthy participants: Between 18 and 65 years | 23 | 42 | 30 | 56 | 406 | 557
    Healthy participants: >=65 years | 0 | 0 | 0 | 0 | 0 | 0
    Anxiety Subjects: number analyzed (Participants) | 78 | 34 | 32 | 34 | 183 | 361
    Anxiety Subjects: <=18 years | 0 | 0 | 0 | 0 | 0 | 0
    Anxiety Subjects: Between 18 and 65 years | 78 | 34 | 32 | 34 | 183 | 361
    Anxiety Subjects: >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Study comprised of several sub-studies with the aim of comparing Healthy participants to Anxiety participants
  Participants
    Healthy Participants: number analyzed (Participants) | 23 | 42 | 30 | 56 | 406 | 557
    Healthy Participants: Female | 13 | 28 | 25 | 43 | 236 | 345
    Healthy Participants: Male | 10 | 14 | 5 | 13 | 170 | 212
    Anxiety Patients: number analyzed (Participants) | 78 | 34 | 32 | 34 | 183 | 361
    Anxiety Patients: Female | 54 | 30 | 28 | 16 | 116 | 244
    Anxiety Patients: Male | 24 | 4 | 4 | 18 | 67 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Study comprised of several sub-studies with the aim of comparing Healthy participants to Anxiety participants
  Participants
    Healthy Participants: number analyzed (Participants) | 23 | 42 | 30 | 56 | 406 | 557
    Healthy Participants: Hispanic or Latino | 2 | 5 | 0 | 6 | 36 | 49
    Healthy Participants: Not Hispanic or Latino | 21 | 36 | 30 | 49 | 359 | 495
    Healthy Participants: Unknown or Not Reported | 0 | 1 | 0 | 1 | 11 | 13
    Anxiety Subjects: number analyzed (Participants) | 78 | 34 | 32 | 34 | 183 | 361
    Anxiety Subjects: Hispanic or Latino | 5 | 6 | 1 | 2 | 20 | 34
    Anxiety Subjects: Not Hispanic or Latino | 71 | 27 | 31 | 32 | 159 | 320
    Anxiety Subjects: Unknown or Not Reported | 2 | 1 | 0 | 0 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Study comprised of several sub-studies with the aim of comparing Healthy participants to Anxiety participants
  Participants
    Healthy Participants: number analyzed (Participants) | 23 | 42 | 30 | 56 | 406 | 557
    Healthy Participants: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 2 | 2
    Healthy Participants: Asian | 5 | 7 | 6 | 5 | 39 | 62
    Healthy Participants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 2 | 2
    Healthy Participants: Black or African American | 7 | 8 | 5 | 20 | 79 | 119
    Healthy Participants: White | 9 | 21 | 17 | 25 | 245 | 317
    Healthy Participants: More than one race | 0 | 3 | 2 | 3 | 10 | 18
    Healthy Participants: Unknown or Not Reported | 2 | 3 | 0 | 3 | 29 | 37
    Anxiety Subjects: number analyzed (Participants) | 78 | 34 | 32 | 34 | 183 | 361
    Anxiety Subjects: American Indian or Alaska Native | 2 | 0 | 0 | 0 | 0 | 2
    Anxiety Subjects: Asian | 7 | 5 | 2 | 2 | 11 | 27
    Anxiety Subjects: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
    Anxiety Subjects: Black or African American | 25 | 8 | 6 | 4 | 36 | 79
    Anxiety Subjects: White | 34 | 17 | 21 | 26 | 110 | 208
    Anxiety Subjects: More than one race | 6 | 3 | 1 | 1 | 6 | 17
    Anxiety Subjects: Unknown or Not Reported | 4 | 1 | 2 | 1 | 19 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent of Correct Button Presses During Threat Compared to the Safe Condition (AAST)
Description: Subjects participated in go/no go (GNG) task condition during periods of threat of shocks and periods of safety when no shock could be administered. During the GNG stimuli were presented on a monitor. In the GNG task, participants were asked to respond to frequent 'go' stimuli ('=') by pressing the '2' on the keypad of a computer keyboard and to withhold their response to infrequent 'nogo' stimuli ('O'). Stimuli were randomly distributed. A correct go hit was a response recorded during these 2000 ms to a go trial. Similarly, a correct nogo omission was a no response during the same period to a nogo trial. Performance was determined for each condition (threat, safe) and trial type (go, nogo) by dividing the number of correct responses by the total number of each trial type. Improvement in accuracy was measured as a higher percent of correct button presses during threat compared to safety.
Time Frame: 2000 ms during trial
Population: Analysis included only participants in sub-study 7 who completed the active avoidance signal task (AAST). Two healthy controls were excluded from analyses.
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Groups:
- Substudy 7/ Active Avoidance Signal Task (AAST) - Healthy Participants; Substudy 7/ Active Avoidance Signal Task (AAST) - Anxiety Patients: Participants performed paradigms which tested whether threat impacts the initiation and the inhibition of behavioral responses
Arm/Group | Substudy 7/ Active Avoidance Signal Task (AAST) - Healthy Participants | Substudy 7/ Active Avoidance Signal Task (AAST) - Anxiety Patients
Number analyzed (Participants) | 22 | 23
Percentage of accurate responses | -0.016 (0.03) | 0.008 (0.04)

2. Primary Outcome: Change in Percent of Correct no Button Presses During Threat Compared to the Safe Condition
Description: as for outcome 1
Time Frame: 2000 ms during trial
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Arm/Group | Substudy 7/ Active Avoidance Signal Task (AAST) - Healthy Participants | Substudy 7/ Active Avoidance Signal Task (AAST) - Anxiety Patients
Number analyzed (Participants) | 22 | 23
Percentage of accurate responses | -0.002 (0.03) | 0.028 (0.04)

3. Primary Outcome: Correct-go Reaction Time (RT) - Safe Condition
Description: Correct go responses were go trials followed by button press. Reaction time (RT) is the time it takes to respond to stimuli. Participants RTs were measured while undergoing alternating periods of safety and shock threat conditions i.e. while anticipating unpleasant electric shocks (threat) or no shock (safe). Mean reaction time (RT) was calculated for correct-go to evaluate speed-accuracy trade-off.
Time Frame: 2000 ms during trial
Population: Analysis included only participants in sub-study 7 who completed the Sustained attention response task (SART).
Measure: Mean (Standard Error); unit: milliseconds (ms)
Groups:
- Substudy 7/ Sustained Attention Response Task (SART) - Healthy Participants; Substudy 7/ Sustained Attention Response Task (SART) - Anxiety Patients: Participants were presented with stimuli and either initiated a response (i.e. "go") or inhibited their response (i.e. "stop") based on what stimuli were presented.
Arm/Group | Substudy 7/ Sustained Attention Response Task (SART) - Healthy Participants | Substudy 7/ Sustained Attention Response Task (SART) - Anxiety Patients
Number analyzed (Participants) | 41 | 41
milliseconds (ms) | 387.8 (16.2) | 337.3 (10.7)

4. Primary Outcome: Correct-go Reaction Time (RT) - Threat Condition
Description: as for outcome 3
Time Frame: 2000 ms during trial
Population: Analysis included only participants in sub-study 7 who completed the Sustained attention response task (SART).
Measure: Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | Substudy 7/ Sustained Attention Response Task (SART) - Healthy Participants | Substudy 7/ Sustained Attention Response Task (SART) - Anxiety Patients
Number analyzed (Participants) | 41 | 41
milliseconds (ms) | 377.4 (14.7) | 332.2 (10.9)

5. Primary Outcome: Go Correct Hits Followed by Button Press - Safe Condition
Description: Subjects participated in go/no go (GNG) task condition during periods of threat of shocks and periods of safety when no shock could be administered. During the GNG stimuli were presented on a monitor. In the GNG task, participants were asked to respond to frequent 'go' stimuli ('=') by pressing the '2' on the keypad of a computer keyboard and to withhold their response to infrequent 'nogo' stimuli ('O'). Stimuli were randomly distributed. A correct go hit was a response recorded during these 2000 ms to a go trial. Similarly, a correct nogo omission was a no response during the same period to a nogo trial. Performance was determined for each condition (threat, safe) and trial type (go, nogo) by dividing the number of correct response by the total number of each trial type.
Time Frame: 2000 ms during trial
Population: Analysis included only participants in sub-study 7 who completed the Sustained attention response task (SART).
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | Substudy 7/ Sustained Attention Response Task (SART) - Healthy Participants | Substudy 7/ Sustained Attention Response Task (SART) - Anxiety Patients
Number analyzed (Participants) | 41 | 41
Proportion of correct responses | 0.91 (0.01) | 0.87 (0.01)

6. Primary Outcome: Go Correct Hits Followed by Button Press - Threat Condition
Description: Subjects participated in go/no go (GNG) task condition during periods of threat of shocks and periods of safety when no shock could be administered. During the GNG stimuli were presented on a monitor. In the GNG task, participants were asked to respond to frequent (91%) 'go' stimuli ('=') by pressing the '2' on the keypad of a computer keyboard and to withhold their response to infrequent (9%) 'nogo' stimuli ('O'). Stimuli were randomly distributed. A correct go hit was a response recorded during these 2000 ms to a go trial. Similarly, a correct nogo omission was a no response during the same period to a nogo trial. Performance was determined for each condition (threat, safe) and trial type (go, nogo) by dividing the number of correct response by the total number of each trial type.
Time Frame: 2000 ms during trial
Population: Analysis included only participants in sub-study 7 who completed the sustained attention response task (SART).
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | Substudy 7/ Sustained Attention Response Task (SART) - Healthy Participants | Substudy 7/ Sustained Attention Response Task (SART) - Anxiety Patients
Number analyzed (Participants) | 41 | 41
Proportion of correct responses | 0.9 (0.01) | 0.87 (0.02)

7. Primary Outcome: Nogo Trials Followed by no Button Press - Safe Condition
Description: as for outcome 5
Time Frame: 2000 ms during trial
Population: Analysis included only participants in sub-study 7 who completed the sustained attention response task (SART).
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | Substudy 7/ Sustained Attention Response Task (SART) - Healthy Participants | Substudy 7/ Sustained Attention Response Task (SART) - Anxiety Patients
Number analyzed (Participants) | 41 | 41
Proportion of correct responses | 0.76 (0.02) | 0.76 (0.01)

8. Primary Outcome: Nogo Trials Followed by no Button Press - Threat Condition
Description: as for outcome 5
Time Frame: 2000 ms during trial
Population: Analysis included only participants in sub-study 7 who completed the sustained attention response task (SART).
Measure: Mean (Standard Error); unit: Proportion of correct responses
Arm/Group | Substudy 7/ Sustained Attention Response Task (SART) - Healthy Participants | Substudy 7/ Sustained Attention Response Task (SART) - Anxiety Patients
Number analyzed (Participants) | 41 | 41
Proportion of correct responses | 0.8 (0.02) | 0.81 (0.02)

9. Primary Outcome: Stroop Effect on Accuracy During Congruent Task Viewing Positive Images: Safe Condition
Description: Participants watched as six trial types differing by congruence and emotion (negative, neutral, positive) were presented during condition blocks (safe, threat) on a computer screen. Each trial began with a fixation point which was then immediately followed by a picture stimulus, followed by a numerical display, followed by a repeat of the picture stimulus, and followed by a blank screen. During threat, a participant could receive a shock. During safe, a participant could not receive a shock. The effect of accuracy on congruence across negative, positive, and neutral images in threat and safe conditions was assessed by participants accurate identification of facial expression.
Time Frame: 11.2 minutes per run for a total of 22.4 minutes
Population: Analysis included only participants in sub-study 5 who completed the face stroop task.
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Groups:
- Substudy 5 /Face Stroop Task - Healthy Participants; Substudy 5 /Face Stroop Task - Anxiety Patients: Stimuli were pictures of faces exhibiting anger, disgust, fear, happiness, sadness and surprise (Ekman, 1993). Intermixed with the faces were pleasant and unpleasant pictures. Subjects indicated which emotion the face displayed. Accurate response was used as measure of facial emotion recognition. Sub-study tested anxiety patients and healthy controls.
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Percentage of accurate responses | 93.9 (0.8) | 95.7 (0.7)

10. Primary Outcome: Stroop Effect on Accuracy During Congruent Task Viewing Positive Images: Threat Condition
Description: as for outcome 9
Time Frame: 11.2 minutes per run for a total of 22.4 minutes
Population: Analysis included only participants in sub-study 5 who completed the face stroop task. Two participants were excluded from the final analysis.
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Percentage of accurate responses | 94.9 (0.9) | 96.0 (0.8)

11. Primary Outcome: Stroop Effect on Accuracy During Congruent Task Viewing Negative Images: Safe Condition
Description: as for outcome 9
Time Frame: 11.2 minutes per run for a total of 22.4 minutes
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Percentage of accurate responses | 94.3 (1.1) | 94.3 (0.8)

12. Primary Outcome: Stroop Effect on Accuracy During Congruent Task Viewing Negative Images: Threat Condition
Description: as for outcome 9
Time Frame: 11.2 minutes per run for a total of 22.4 minutes
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Percentage of accurate responses | 95.3 (0.7) | 95.9 (0.8)

13. Primary Outcome: Stroop Effect on Accuracy During Congruent Task Viewing Neutral Images: Safe Condition
Description: as for outcome 9
Time Frame: 11.2 minutes per run for a total of 22.4 minutes
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Percentage of accurate responses | 94.9 (0.8) | 95.1 (0.8)

14. Primary Outcome: Stroop Effect on Accuracy During Congruent Task Viewing Neutral Images: Threat Condition
Description: as for outcome 9
Time Frame: 11.2 minutes per run for a total of 22.4 minutes
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Percentage of accurate responses | 96.2 (0.8) | 96.7 (0.5)

15. Primary Outcome: Stroop Effect on Accuracy During Incongruent Task Viewing Positive Images: Safe Condition
Description: as for outcome 9
Time Frame: 11.2 minutes per run for a total of 22.4 minutes
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Percentage of accurate responses | 94.1 (1) | 96.5 (0.6)

16. Primary Outcome: Stroop Effect on Accuracy During Incongruent Task Viewing Positive Images: Threat Condition
Description: as for outcome 9
Time Frame: 11.2 minutes per run for a total of 22.4 minutes
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Percentage of accurate responses | 94.3 (0.9) | 94.1 (1)

17. Primary Outcome: Stroop Effect on Accuracy During Incongruent Task Viewing Negative Images: Safe Condition
Description: as for outcome 9
Time Frame: 11.2 minutes per run for a total of 22.4 minutes
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Percentage of accurate responses | 94.2 (0.9) | 94.0 (0.7)

18. Primary Outcome: Stroop Effect on Accuracy During Incongruent Task Viewing Negative Images: Threat Condition
Description: as for outcome 9
Time Frame: 11.2 minutes per run for a total of 22.4 minutes
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Percentage of accurate responses | 95.0 (0.7) | 95.3 (0.8)

19. Primary Outcome: Stroop Effect on Accuracy During Incongruent Task Viewing Neutral Images: Safe Condition
Description: as for outcome 9
Time Frame: 11.2 minutes per run for a total of 22.4 minutes
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Percentage of accurate responses | 94.4 (1.1) | 94.8 (0.7)

20. Primary Outcome: Stroop Effect on Accuracy During Incongruent Task Viewing Neutral Images: Threat Condition
Description: as for outcome 9
Time Frame: 11.2 minutes per run for a total of 22.4 minutes
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Percentage of accurate responses
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Percentage of accurate responses | 95.8 (0.7) | 95.8 (0.7)

21. Primary Outcome: Subjective Rating of Difficulty With Attention During Safe Condition
Description: Following tasks completion, participants provided retrospective ratings of: anxiety and attention during safe and threat conditions using an analog scale ranging from 1 (not at all) to 10 (extremely). Participants rated overall subjective difficulty with attention ('How difficult was it to pay attention during threat/safe?') and level of anxiety ('How anxious were you during threat/safe?'). Retrospective ratings of anxiety and difficulty with attention were analyzed with two way Diagnosis x Condition (safe, threat) ANOVA.
Time Frame: Assessed immediately after completing the affective Stroop task
Population: as for outcome 10
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
units on a scale | 2.9 (0.4) | 4.1 (0.4)

22. Primary Outcome: Subjective Rating of Difficulty With Attention During Threat Condition
Description: as for outcome 21
Time Frame: Assessed immediately after completing the affective Stroop task
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Units on a scale | 4.4 (0.5) | 6.5 (0.4)

23. Primary Outcome: Subjective Rating of Level of Anxiety During Safe Condition
Description: as for outcome 21
Time Frame: Assessed immediately after completing the affective Stroop task
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Units on a scale | 2 (0.3) | 3.5 (0.4)

24. Primary Outcome: Subjective Rating of Level of Anxiety During Threat Condition
Description: as for outcome 21
Time Frame: Assessed immediately after completing the affective Stroop task
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Substudy 5 /Face Stroop Task - Healthy Participants | Substudy 5 /Face Stroop Task - Anxiety Patients
Number analyzed (Participants) | 31 | 36
Units on a scale | 6.7 (0.5) | 8.1 (0.3)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Substudy 1/ Neutral, Predictable, and Unpredictable Responses - Healthy Participants; Substudy 1/ Neutral, Predictable, and Unpredictable Responses - Anxiety Subjects: This experiment examined physiological responses including startle reflex to different threat of shock conditions (neutral (N)- no shock, unpredictable - shock at any time , and predictable -cued shock (P)) in subjects with anxiety disorders and healthy control. Each of these conditions were signaled by a written text displayed on a computer monitor (e.g., shock only when blue square present).
- Substudy 2/Working Memory Task - Healthy Participants; Substudy 2/Working Memory Task - Anxiety Subjects: Subjects performed a working memory task in two conditions, under threat of shock and in safety (no threat of shock). Subjects included participants with anxiety disorder and healthy volunteer.
- Substudy 5/Face Stroop Task - Healthy Participants; Substudy 5/Face Stroop Task - Anxiety Subjects: Stimuli were pictures of faces exhibiting anger, disgust, fear, happiness, sadness and surprise. Intermixed with the faces were pleasant, unpleasant, and neutral pictures. Subjects indicated which emotion the face displayed. Accurate response was used as measure of facial emotion recognition. Subjects included participants with anxiety disorder and healthy volunteer.
- Substudy 7/Active Avoidance and Sustained Attention Tasks - Healthy Participants; Substudy 7/Active Avoidance and Sustained Attention Tasks - Anxiety Subjects: In the active avoidance signal task (AAST), participants performed paradigms which tested whether threat impacts the initiation and the inhibition of behavioral responses. In the sustained attention response task (SART), participants were presented with stimuli and either initiated a response (i.e. "go") or inhibited their response (i.e. "stop") based on what stimuli were presented. Subjects included participants with anxiety disorder and healthy volunteer.
- Pilot Tasks - Healthy Participants; Pilot Tasks - Anxiety Subjects: Participants completed one or more pilot tasks: nerve stimulation, short speech in front of a small audience or in a virtual environment, burst of air to neck, provide saliva samples for cortisol analysis, squeeze a grip device, virtual reality task, and/or computer based experimental tasks.
Arm/Group | Substudy 1/ Neutral, Predictable, and Unpredictable Responses - Healthy Participants | Substudy 1/ Neutral, Predictable, and Unpredictable Responses - Anxiety Subjects | Substudy 2/Working Memory Task - Healthy Participants | Substudy 2/Working Memory Task - Anxiety Subjects | Substudy 5/Face Stroop Task - Healthy Participants | Substudy 5/Face Stroop Task - Anxiety Subjects | Substudy 7/Active Avoidance and Sustained Attention Tasks - Healthy Participants | Substudy 7/Active Avoidance and Sustained Attention Tasks - Anxiety Subjects | Pilot Tasks - Healthy Participants | Pilot Tasks - Anxiety Subjects
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/78 | 0/42 | 0/35 | 0/33 | 0/36 | 0/65 | 0/91 | 0/406 | 0/183
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/78 | 0/42 | 0/35 | 0/33 | 0/36 | 0/65 | 0/91 | 0/406 | 0/183
Other Adverse Events (participants affected / at risk) | 0/23 | 0/78 | 0/42 | 0/35 | 0/33 | 0/36 | 0/65 | 0/91 | 0/406 | 0/183

LIMITATIONS AND CAVEATS:
This protocol was a series of sub-studies using sample subjects which explains the low numbers of participants per study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT00055224/Prot_SAP_000.pdf